CLINICAL TRIAL: NCT07151417
Title: Adjunctive Use of Corticosteroid in Periarticular Injections in Primary Total Knee Arthroplasty
Brief Title: Use of Corticosteroid in Intraopertive Injections in Total Knee Replacement Surgery.
Acronym: TKACSI
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ian P. Marshall, Resident Physician, Orthopaedic Surgery, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-21385
Record Dates: First submitted 2025-08-13; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Musculoskeletal Disease; Surgery
Keywords: total knee arthroplasty (TKA); manipulation under anesthesia (MUA); corticosteroid; periarticular injection/pericapsular injection (PAI); zilretta
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Diseases | interventions — Steroids; Methylprednisolone; Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Masking Description: Research participants will be randomized to one of three groups unless they are diabetic or pre-diabetic then they will be randomized to one of 2 groups (Group 1 or Group 3). Participants will not know to which group they were randomized to.
  The groups that participants will be randomized to are:
  Group 1: Standard PAI: 30 mg Toradol/ketorolac (30mg/ml), 49.25ml 0.5% ropivacaine (5mg/ml), and 0.5 mg epinephrine (1mg/ml), 0.8 ml clonidine (0.1mg/ml) and 8.45 ml 0.9% sodium chloride Group 2: Standard PAI + 40mg methylprednisolone (diabetics and pre-diabetics will not be randomized to this group) Group 3: Standard PAI + 32mg Zilretta (triamcinolone acetonide extended release injectable suspension)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard PAI (Active Comparator): Group1 (n=80; 40 non-diabetic and 40 diabetic participants): Standard PAI: 30 mg Toradol/ketorolac (30mg/ml), 49.25ml 0.5% ropivacaine (5mg/ml), and 0.5 mg epinephrine (1mg/ml), 0.8 ml clonidine (0.1mg/ml) and 8.45 ml 0.9% sodium chloride
  Interventions: Drug: PAI
- Methylprednisolone (Active Comparator): 2. Group2 (n=40, non-diabetic): Standard PAI + 40mg methylprednisolone (n = 40)
  Interventions: Drug: PAI + steroid
- Zilretta (Active Comparator): 3. Group3 (n=80; 40 non-diabetic and 40 diabetic participants): Standard PAI + 32mg Zilretta (triamcinolone acetonide extended release injectable suspension)
  Interventions: Drug: PAI + zilretta

INTERVENTIONS:
Drug: PAI — Standard PAI: 30 mg Toradol/ketorolac (30mg/ml), 49.25ml 0.5% ropivacaine (5mg/ml), and 0.5 mg
  Arms: Standard PAI
Drug: PAI + steroid — Standard PAI + 40mg methylprednisolone (n = 40)
  Other Names: PAI + methylprednisolone
  Arms: Methylprednisolone
Drug: PAI + zilretta — Standard PAI + 32mg Zilretta (triamcinolone acetonide extended release injectable suspension)
  Arms: Zilretta

SUMMARY:
The goal of this clinical trial is to find out which type of steroid medicine, when added to a standard pain-control injection during total knee replacement surgery, works best at reducing pain, limiting opioid use, and improving recovery in adults undergoing surgery for severe knee arthritis or injury.

The main questions it aims to answer are:

Does adding a steroid to the injection improve pain control and reduce opioid use after surgery? Is the newer extended-release steroid (Zilretta) more effective and safer-especially for patients with diabetes-than the traditional steroid (methylprednisolone)?

Researchers will compare:

Standard pain-control injection alone Standard injection plus methylprednisolone Standard injection plus Zilretta to see which option provides better pain relief, less opioid use, and improved knee function.

(Patients with diabetes or prediabetes will only be in the standard injection or Zilretta groups so researchers can study whether Zilretta is safer for blood sugar control.)

Participants will:

Be randomly assigned to one of the study groups during their total knee replacement surgery Receive the assigned pain-control injection around the knee joint

Be followed after surgery to measure:

Pain levels Opioid pain medication use Knee movement (range of motion) Whether another procedure (such as manipulation under anesthesia) is needed if the knee becomes too stiff Patient-reported outcome surveys about pain and function

DETAILED DESCRIPTION:
Total knee replacement surgery (also called total knee arthroplasty, or TKA) is a common procedure for people with severe knee arthritis or injury. While the surgery often leads to significant pain relief and improved mobility, the days and weeks afterward can be uncomfortable. Managing pain during recovery is important-not just to make patients feel better, but also to help them move their knee sooner, avoid excessive use of opioid medications, and get back to normal activities faster.

One common pain management tool is called a pericapsular injection (PAI). This is a mixture of medications injected around the knee joint during surgery to help control pain after the operation. PAIs usually include a long-lasting numbing medicine, an anti-inflammatory drug, and sometimes other medications that improve pain relief. Corticosteroids-powerful anti-inflammatory drugs-are sometimes added, but the best type of steroid and the ideal way to give it is still debated among doctors.

Why This Study Is Being Done This study will compare two types of corticosteroids, methylprednisolone (a traditional steroid) and Zilretta (a newer, extended-release form of the steroid triamcinolone), to see which works better when added to the standard PAI. Zilretta releases medication slowly over time, which may lead to longer-lasting pain control and fewer side effects such as temporary increases in blood sugar-something especially important for people with diabetes.

How the Study Works

Patients having total knee replacement will be randomly placed into one of three groups:

1. Standard PAI only - This mixture includes a long-acting numbing medicine, an anti-inflammatory (ketorolac), a small dose of adrenaline (epinephrine), clonidine (to help with pain control), and sterile saline.
2. Standard PAI + methylprednisolone - The same standard mixture with the addition of 40 mg of methylprednisolone.
3. Standard PAI + Zilretta - The same standard mixture with 32 mg of Zilretta, the extended-release steroid.

People with diabetes or prediabetes will only be placed in groups 1 or 3 so researchers can compare how Zilretta affects them compared to no steroid at all.

What Will Be Measured

The researchers will check patients' progress at several points after surgery to investigate:

* Pain levels
* Opioid pain medication use (measured in morphine-equivalent doses)
* Knee movement (range of motion)
* Need for further procedures (such as manipulation under anesthesia, or MUA, if the knee becomes too stiff)
* Patient-reported outcome surveys (including the Knee Injury and Osteoarthritis Outcome Score and the Single Assessment Numeric Evaluation) Expected Findings

The team believes that adding a corticosteroid to the PAI will:

* Improve pain control
* Reduce the need for opioid medications
* Lower the risk of needing a manipulation procedure to improve range of motion They also expect that Zilretta, because it lasts longer, will work better than methylprednisolone-especially in people with diabetes, by offering pain relief without causing as much temporary increase in blood sugar.

Why This Matters Past research shows that PAIs can help reduce pain and the need for opioids after knee replacement surgery, without raising the risk of infection or other serious complications. But doctors still don't know which steroid is best to use. If Zilretta works better and causes fewer side effects, it could become the preferred option for many patients-particularly those with other health issues like diabetes.

The results of this study could help guide surgeons toward the safest and most effective pain control strategies for people recovering from knee replacement surgery, ultimately leading to better recoveries, fewer complications, and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients within the MHS who are DEERS eligible undergoing primary TKA at Walter Reed National Military Medical Center (WRNMMC), Surgery Center of Chevy Chase or District Surgery Center
* Age 18 or older
* successful surgical intervention

Exclusion Criteria:

* Unicompartmental knee arthroplasty (UKA)
* Revision total knee arthroplasty (rTKA)
* Females who are pregnant or nursing
* Allergic to ingredients in PAI or previous adverse reaction to steroids being used in this study
* Diabetics will be excluded from Group 2 (standard PAI + methylprednisolone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to determine whether total knee arthroplasty outcomes are significantly better for Zilretta (Group 3) and methylprednisolone (Group 2) as compared to standard PAI (Group 1) and Zilretta versus methylprednisolone. | 24 hours, 72 hours, 7 days, and 28 days post
  The following outcomes after total knee arthroplasty will be compared to determine whether outcomes are significantly better for Zilretta (Group 3) and methylprednisolone (Group 2) as compared to standard PAI (Group 1) and Zilretta versus methylprednisolone:
  • Improvement in pain levels postoperatively based on measurement of pain intensity using a Visual Analogue Scale (VAS) at 24hrs, 72 hours, and 7 days (all phone call), and 28 days
Postoperative ROM | 28, 120 and 365 days postop
  The following outcomes after total knee arthroplasty will be compared to determine whether outcomes are significantly better for Zilretta (Group 3) and methylprednisolone (Group 2) as compared to standard PAI (Group 1) and Zilretta versus methylprednisolone: Change in range of motion (ROM) at 28, 120 and 365 days postop
Patient reported outcome measure | 120 and 365 days postoperatively
  The following outcomes after total knee arthroplasty will be compared to determine whether outcomes are significantly better for Zilretta (Group 3) and methylprednisolone (Group 2) as compared to standard PAI (Group 1) and Zilretta versus methylprednisolone:
  • Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) score at 120 and 365 days postoperatively
Patient reported outcome measures 2 | 120 and 365 days postop
  The following outcomes after total knee arthroplasty will be compared to determine whether outcomes are significantly better for Zilretta (Group 3) and methylprednisolone (Group 2) as compared to standard PAI (Group 1) and Zilretta versus methylprednisolone:
  • Change in Single Assessment Numeric Evaluation (SANE) score at 120 and 365 days postop
Postop pain medication usage | 24hrs, 72 hours, and 7 days, and 28 days postop
  The following outcomes after total knee arthroplasty will be compared to determine whether outcomes are significantly better for Zilretta (Group 3) and methylprednisolone (Group 2) as compared to standard PAI (Group 1) and Zilretta versus methylprednisolone:
  • Decreased morphine equivalent (MEQ) postoperatively at 24hrs, 72 hours, and 7 days (all phone call), and 28 days
MUA rate | 28 days postop
  The following outcome after total knee arthroplasty will be compared to determine whether outcomes are significantly better for Zilretta (Group 3) and methylprednisolone (Group 2) as compared to standard PAI (Group 1) and Zilretta versus methylprednisolone:
  • Decreased manipulation under anesthesia rates (MUA) compared to historical rate at our institution at 28 days

SECONDARY OUTCOMES:
Adverse events and subgroup analysis | 28 days, 120 days, 365 days postop
  To determine whether the adverse event rates associated with Zilretta and methylprednisolone are significantly less than the adverse event rates for standard PAI.

CONTACTS AND LOCATIONS:
Overall Officials: John P Cody, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Li Z, Gao X, Lin J. The efficacy and safety of intra-articular injection of corticosteroids in multimodal analgesic cocktails in total knee arthroplasty-a historically controlled study. Front Surg. 2024 Jun 11;11:1279462. doi: 10.3389/fsurg.2024.1279462. eCollection 2024. PMID 38919978
- [Background] Wainwright JD, Gugala Z, Krueger CA, Wenke JC. Adding corticosteroids to intra-operative periarticular injections in total knee arthroplasty: A systematic review. Knee. 2024 Aug;49:87-96. doi: 10.1016/j.knee.2024.05.009. Epub 2024 Jun 13. PMID 38876084
- [Background] Wainwright JD, Alaraj S, Wenke JC. Systematic review of intraoperative corticosteroid injections and the risk of infection in arthroscopic surgery. J Clin Orthop Trauma. 2024 Jan 3;48:102332. doi: 10.1016/j.jcot.2024.102332. eCollection 2024 Jan. PMID 38282804
- [Background] Su C, Liu Y, Wu P, Lang J, Chen L. Comparison Between Periarticular Analgesia Versus Intraarticular Injection for Effectiveness and Safety After Total Knee Arthroplasty. J Perianesth Nurs. 2022 Dec;37(6):952-955. doi: 10.1016/j.jopan.2022.04.010. Epub 2022 Sep 16. PMID 36123240
- [Background] Sreedharan Nair V, Ganeshan Radhamony N, Rajendra R, Mishra R. Effectiveness of intraoperative periarticular cocktail injection for pain control and knee motion recovery after total knee replacement. Arthroplast Today. 2019 Jul 12;5(3):320-324. doi: 10.1016/j.artd.2019.05.004. eCollection 2019 Sep. PMID 31516975
- [Background] Schwartz A, Cochrane NH, Jiranek WA, Ryan SP. Periarticular Injection in Total Knee Arthroplasty. J Am Acad Orthop Surg. 2023 Jun 15;31(12):614-619. doi: 10.5435/JAAOS-D-22-01179. Epub 2023 Apr 14. PMID 37071876
- [Background] Russell SJ, Sala R, Conaghan PG, Habib G, Vo Q, Manning R, Kivitz A, Davis Y, Lufkin J, Johnson JR, Kelley S, Bodick N. Triamcinolone acetonide extended-release in patients with osteoarthritis and type 2 diabetes: a randomized, phase 2 study. Rheumatology (Oxford). 2018 Dec 1;57(12):2235-2241. doi: 10.1093/rheumatology/key265. PMID 30203101
- [Background] Oshima A, Hatayama K, Terauchi M, Kakiage H, Hashimoto S, Chikuda H. The comparison of dexamethasone and triamcinolone periarticular administration in total knee arthroplasty: retrospective cohort study. BMC Musculoskelet Disord. 2022 Feb 5;23(1):120. doi: 10.1186/s12891-022-05048-8. PMID 35123474
- [Background] Moon HK, Han CD, Yang IH, Cha BS. Factors affecting outcome after total knee arthroplasty in patients with diabetes mellitus. Yonsei Med J. 2008 Feb 29;49(1):129-37. doi: 10.3349/ymj.2008.49.1.129. PMID 18306479
- [Background] Liu M, Zhang D, Shi B. Comparison of the Post-Total Knee Arthroplasty Analgesic Effect of Intraoperative Periarticular Injection of Different Analgesics. J Coll Physicians Surg Pak. 2019 Dec;29(12):1169-1172. doi: 10.29271/jcpsp.2019.12.1169. PMID 31839089
- [Background] Li Q, Mu G, Liu X, Chen M. Efficacy of additional corticosteroids to multimodal cocktail periarticular injection in total knee arthroplasty: a meta-analysis of randomized controlled trials. J Orthop Surg Res. 2021 Jan 22;16(1):77. doi: 10.1186/s13018-020-02144-0. PMID 33482865
- [Background] Kulkarni M, Mallesh M, Wakankar H, Prajapati R, Pandit H. Effect of Methylprednisolone in Periarticular Infiltration for Primary Total Knee Arthroplasty on Pain and Rehabilitation. J Arthroplasty. 2019 Aug;34(8):1646-1649. doi: 10.1016/j.arth.2019.04.060. Epub 2019 May 2. PMID 31155459
- [Background] Kim JI, Kim YT, Jung HJ, Lee JK. Does adding corticosteroids to periarticular injection affect the postoperative acute phase response after total knee arthroplasty? Knee. 2020 Mar;27(2):493-499. doi: 10.1016/j.knee.2019.10.029. Epub 2019 Dec 2. PMID 31806506
- [Background] Kim DH, Beathe JC, Lin Y, YaDeau JT, Maalouf DB, Goytizolo E, Garnett C, Ranawat AS, Su EP, Mayman DJ, Memtsoudis SG. Addition of Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee and Adductor Canal Block to Periarticular Injection Enhances Postoperative Pain Control in Total Knee Arthroplasty: A Randomized Controlled Trial. Anesth Analg. 2019 Aug;129(2):526-535. doi: 10.1213/ANE.0000000000003794. PMID 30234517
- [Background] Kg G, J R. Efficacy of Intraoperative Periarticular Local Infiltration for Pain Control and Ambulation in Total Knee Arthroplasty: A Randomized Case-Control Study. Cureus. 2024 Jan 20;16(1):e52639. doi: 10.7759/cureus.52639. eCollection 2024 Jan. PMID 38380215
- [Background] Hannon CP, Fillingham YA, Spangehl MJ, Karas V, Kamath AF, Casambre FD, Verity TJ, Nelson N, Hamilton WG, Della Valle CJ. The Efficacy and Safety of Periarticular Injection in Total Joint Arthroplasty: A Direct Meta-Analysis. J Arthroplasty. 2022 Oct;37(10):1928-1938.e9. doi: 10.1016/j.arth.2022.03.045. PMID 36162925